CLINICAL TRIAL: NCT05366348
Title: Investigation of the Effects of Horse-back Riding on Core Muscles in Adolescents
Brief Title: The Effects of Horse-back Riding on Core Muscles in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pınar Kuyulu (Other)
Responsible Party: Sponsor-Investigator, Pınar Kuyulu, Director, Sanko University
Organization: Sanko University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/01-40
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Health, Subjective; Activity, Motor; Muscle Strength
Keywords: Balance; Core stability; Adolescent; muscle strength; horseback riding
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horse-back riding (Experimental): The study group received horse-back riding training for eight weeks.
  Interventions: Other: Recreational activity
- Control group (No Intervention): Sedentary adolescent individuals who do not ride horses

INTERVENTIONS:
Other: Recreational activity — Horse-back riding
  Arms: Horse-back riding

SUMMARY:
The aim of the study is to examine the effects of riding on the core muscles, balance and muscle strength of the extremities in healthy adolescents.

Core strength, core endurance, balance, upper extremity and lower extremity strength assessments were performed on the study group before and after the riding training.

DETAILED DESCRIPTION:
Twenty participants, aged between 10-19 years, research (n=10) and control (n=10) groups, were included in the study. The study group (n=10) received riding training for eight weeks. The study group was evaluated twice before and after riding.The control group only participated in the assessments at the start of the study. Demographic information of all volunteer participants were recorded.

Core strength was evaluated with a stabilizer pressure biofeedback device, and core endurance was evaluated with isometric endurance tests. Balance was evaluated with Star Excursion Balance Test, upper extremity strength was evaluated with hand dynamometer and lower extremity strength was evaluated with back-leg dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 10-19 years
* No previous horse-back riding experience
* Individuals with no health problems

Exclusion Criteria

* Any history of surgery intervention
* Individuals who do not regularly participate in horse-back riding

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Core stability | 8 weeks
  Core strength was measured with a stabilizer pressure biofeedback device. Core endurance was evaluated with isometric endurance tests.

SECONDARY OUTCOMES:
Balance | 8 weeks
  Star excursion balance test
Extremity strength | 8 weeks
  Hand dynamometer and Back&leg dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kuyulu, MsC(c), Study Director — Sanko University
Locations (1):
- SANKO University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No